CLINICAL TRIAL: NCT02624323
Title: Real-time Ultrasound-guided Axillary and Jugular Vein Catheterization: A Prospective Comparison in Mechanically Ventilated Critically Ill Patients. A Randomized Study
Brief Title: Ultrasound Guided Axillary Versus Jugular Central Venous Catheterization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniwersytecki Szpital Kliniczny w Opolu (Other)
Responsible Party: Principal Investigator, Tomasz Czarnik, MD PhD, Principal Investigator, Uniwersytecki Szpital Kliniczny w Opolu
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AxillaryJugularUSG-RCT
Record Dates: First submitted 2015-11-29; First posted 2015-12-08 (Estimated); Last update posted 2020-08-04 (Actual); Status verified 2020-08

CONDITIONS: Critical Illness
Keywords: ultrasonography; catheterization; central line; mechanical ventilation; intensive care; axillary vein; jugular vein; randomization
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Axillary catheterization (Experimental): Real-time ultrasound-guided axillary vein catheterization, in plain technique.
  Interventions: Procedure: Real-time ultrasound-guided central vein catheterization.
- Jugular catheterization (Experimental): Real-time ultrasound-guided jugular vein catheterization, out of plain technique.
  Interventions: Procedure: Real-time ultrasound-guided central vein catheterization.

INTERVENTIONS:
Procedure: Real-time ultrasound-guided central vein catheterization.

SUMMARY:
The main intention of this study is to compare two ultrasound-guided central venous catheterization procedures namely: real-time, ultrasound-guided, in plane axillary vein catheterization and real-time, ultrasound-guided, out of plane jugular vein catheterization in terms of venipuncture, catheterization success, early mechanical complication and catheter-related infection rate in mechanically ventilated patients admitted to the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* mechanically ventilated intensive care patients with clinical indications for central venous line placement

Exclusion Criteria:

* trauma and hematoma at the catheterization site
* major blood coagulation disorders coincided with active bleeding
* anatomical abnormalities at the catheterization site
* infection at the catheterization site
* age less than 18 years
* lack of patients or closest relatives consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 614 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Procedure success rate | 24 hours
  to define catheterization success rate

SECONDARY OUTCOMES:
Incidence of Catheter colonization | 1 month
  to assess the incidence of catheter colonization after removal
Incidence of catheter-related bloodstream infection | 1 month
  to assess the incidence of catheter-related bloodstream infection
Procedure complication rate | 24 hours
  to assess the early mechanical complication rate

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Czarnik, MD PhD, Principal Investigator — Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu
Locations (2):
- Poland (2):
  - Department of Anesthesiology and Intensive Care, Uniwersytecki Szpital Kliniczny w Opolu, Opole, Silesian Voivodeship
  - 2nd Department of Anesthesiology and Critical Care, Medical University of Lublin, Lublin

REFERENCES:
- [Derived] Czarnik T, Czuczwar M, Borys M, Chrzan O, Filipiak K, Maj M, Marszalski M, Miodonska M, Molsa M, Pietka M, Piwoda M, Piwowarczyk P, Rogalska Z, Stachowicz J, Gawda R. Ultrasound-Guided Infraclavicular Axillary Vein Versus Internal Jugular Vein Cannulation in Critically Ill Mechanically Ventilated Patients: A Randomized Trial. Crit Care Med. 2023 Feb 1;51(2):e37-e44. doi: 10.1097/CCM.0000000000005740. Epub 2022 Dec 7. PMID 36476809